CLINICAL TRIAL: NCT01539395
Title: A Cross-Sectional Study of MSDx Complex 1 as a Marker for Active Disease in Multiple Sclerosis
Status: Withdrawn | Type: Observational
Sponsor: MSDx, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: MSDX0211
Record Dates: First submitted 2012-02-21; First posted 2012-02-27 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Multiple Sclerosis
Keywords: Relapsing Remitting; MS
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood remaining after testing for MSDx Complex-1 will be retained for evaluation for other MS biomarkers
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Inactive Disease: Inactive disease; RRMS patients who have been treated with monthly infusions of Tysabri for 12 months and have had stable disease for the last 6 months or more and show stable or improving neurological deficits over 3 months on Tysabri.
  Interventions: Other: MSDx Complex-1 Biomarker Test
- Active Disease: Active disease; RRMS patients in acute clinical relapse or with active MRI. Blood sample obtained within 30 days of event AND before steroid treatment (or) patients in early disease on or off first line agents with relapse in prior 3 months AND not treated with steroids for at least 2 months.
  Interventions: Other: MSDx Complex-1 Biomarker Test
- Active Disease - Steroid Therapy: Patient with a diagnosis of relapsing remitting multiple sclerosis (RRMS) who is about to begin steroid therapy for a relapse in clinical symptoms (either diagnosed clinically or via gadolinium MRI).
  Interventions: Other: MSDx Complex-1 Biomarker Test

INTERVENTIONS:
Other: MSDx Complex-1 Biomarker Test — A biomarker test for the level of MSDx Complex-1

SUMMARY:
This is a Cross-Sectional Study of MSDx Complex 1 as a Marker for Active Disease in Multiple Sclerosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age 45 years or older of either gender and of any racial/ethnic group.
2. Subjects must be in generally good health.
3. Subjects must be able and willing to comply with the requirements of the protocol.
4. Must be diagnosed with RRMS
5. Meets the criteria to enter Group 1 or Group 2

Exclusion Criteria:

1. Subject is currently in middle of an active episode of an autoimmune condition (e.g. rheumatoid arthritis, system lupus erythematosis)
2. Subject currently has a condition such as active influenza that would stimulate the immune system

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who currently diagnosed with relapsing remitting multiple sclerosis
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2012-04 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Biomarker Differential | Baseline
  A difference in the levels of Complex-1 between subjects with controlled, stable MS vs. subjects in acute MS relapse

SECONDARY OUTCOMES:
Biomarker reduction with steroid therapy | 3 months
  A decrease in the level of MSDx Complex-1 in response to steroid therapy for a relapse of MS.

CONTACTS AND LOCATIONS:
Overall Officials: Jeanette K Wendt, MD, Principal Investigator — Northwest NeuroSpecialists, PLLC
Locations (1):
- Northwest NeuroSpecialists, PLLC, Tucson, Arizona, United States